CLINICAL TRIAL: NCT00372723
Title: Pilot Study Comparing Remicade (Infliximab) vs. Standard Care in the Treatment of Toxic Epidermal Necrolysis
Brief Title: Study of a Potential New Treatment for Patients With Toxic Epidermal Necrolysis (TEN)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108983
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Toxic Epidermal Necrolysis
Keywords: toxic epidermal necrlysis; ten
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Infliximab

INTERVENTIONS:
Drug: Remicaide (infliximab) — a single dose infusion of 5mg/kg Remicade (Infliximab)

SUMMARY:
To determine whether treatment of patients who have toxic epidermal necrolysis with a drug called remicaide increases the number of patients who are alive 30 days laters.

DETAILED DESCRIPTION:
This is a pilot (preliminary) study. Patients with a diagnosis of TEN will be asked to consider participating. The study intervention is a single intravenous dose of remicaide (5 mg/kg). Standard supportive care will be given. The percentage of patients alive at 30 days after treatment with remicaide will be compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Admission to burn unit with a histologic diagnosis of TENs

Exclusion Criteria:

* Pregnancy
* hypersensitivity to remicaide
* history of heart failure
* documented bacteremia
* history of cancer
* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
30 day mortality | 30 days

SECONDARY OUTCOMES:
Safety labs and adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gamelli, MD, Principal Investigator — Loyola University Medical Center, Department of Surgery